CLINICAL TRIAL: NCT07096193
Title: Phase 1/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of GS-4321 in Healthy Participants and Participants With Chronic Hepatitis Delta
Brief Title: Study of GS-4321 in Healthy Participants and Participants With Chronic Hepatitis Delta Virus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-567-6968; 2025-522729-36 (Other: EU CT Number)
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis Delta
MeSH Terms: conditions — Hepatitis D, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1: GS-4321 (Experimental): Participants will receive single escalating doses of GS-4321.
  Interventions: Drug: GS-4321
- Phase 1: Placebo (Placebo Comparator): Participants will receive placebo to match the single escalating doses of GS-4321
  Interventions: Drug: GS-4321 Placebo
- Phase 2: GS-4321 (Experimental): Participants will receive multiple escalating doses of GS-4321 up to 96 weeks.
  Interventions: Drug: GS-4321

INTERVENTIONS:
Drug: GS-4321 — Administered subcutaneous (SC) or intravenously IV
  Arms: Phase 1: GS-4321
Drug: GS-4321 Placebo — Administered SC
  Arms: Phase 1: Placebo
Drug: GS-4321 — Administered SC
  Arms: Phase 2: GS-4321

SUMMARY:
The goals of this clinical study are to first learn more about safety and dosing of the study drug GS-4321 in healthy participants. The study will then learn about the safety and effectiveness of GS-4321 in participants with chronic hepatitis delta (CHD).

The primary objective of Phase 1 of this study is to evaluate the safety, tolerability and Pharmacokinetics (PK) of the escalating single doses of GS-4321 administered in healthy participants.

The primary objective of Phase 2 of this study is to evaluate the efficacy and safety of the multiple escalating doses of GS-4321 in participants with CHD.

ELIGIBILITY:
Key Inclusion Criteria:

Part A:

* Participants assigned male or female at birth who are of childbearing potential and engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.
* Have a body mass index (BMI) of ≤ 30.0 kg/m2 at screening and at admission.

Part B:

* Participants assigned male or female at birth who are of childbearing potential and engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.
* Chronic hepatitis delta (CHD) for ≥ 6 months prior to screening, documented by prior medical history.
* Must be receiving a commercially available entecavir, TAF, or TDF for the treatment of hepatitis B virus (HBV) infection at or prior to enrollment. Coformulation as part of a fixed-dose combination for the treatment of HIV is permitted.
* Non-cirrhotic or compensated cirrhosis.
* Hepatitis delta virus ribonucleic acid (HDV RNA ) > 100 IU/mL at screening.
* Alanine aminotransferase (ALT) level > 1 × Upper limit of normal (ULN), but < 10 × ULN at screening.

Key Exclusion Criteria:

Part A:

* Positive serum or urine pregnancy test.
* Participants with plans to breastfeed during the study period.

Part B:

* Positive serum or urine pregnancy test.
* Participants with plans to breastfeed during the study period.
* Current or previous clinically decompensated liver disease, including coagulopathy, hepatic encephalopathy, and esophageal varices hemorrhage due to HDV or HBV.
* Child-Turcotte-Pugh (CTP)-B or -C or a CTP score of ≥ 7.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Phase 1 and 2: Percentage of Participants With Treatment-emergent Adverse Events | Phase 1: First dose up to 44 weeks; Phase 2: First dose up to 96 Weeks plus 48 weeks of posttreatment follow-up
Phase 1 and 2: Percentage of Participants With Treatment-emergent Serious Adverse Events | Phase 1: First dose up to 44 weeks; Phase 2: First dose up to 96 Weeks plus 48 weeks of posttreatment follow-up
Phase 1 and 2: Percentage of Participants Experiencing Treatment-emergent Clinical Laboratory Abnormalities | Phase 1: First dose up to 44 weeks; Phase 2: First dose up to 96 Weeks plus 48 weeks of posttreatment follow-up
Phase 1: Serum Pharmacokinetic (PK) parameter; AUClast of GS-4321 | First dose up to 24 Weeks
  AUClast is defined as the area under the concentration versus time curve from time zero to the last quantifiable concentration.
Phase 1: Serum PK Parameter: AUCinf | First dose up to 24 Weeks
  AUCinf is defined as the area under the concentration versus time curve extrapolated to infinite time.
Phase 1: Serum PK Parameter: Cmax | First dose up to 24 Weeks
  Cmax is defined as the maximum observed concentration of drug.
Phase 1: Serum PK Parameter: Tmax | First dose up to 24 Weeks
  Tmax is defined as the time (observed time point) of Cmax.
Phase 1: Serum PK Parameter: t1/2 | First dose up to 24 Weeks
Phase 2: Proportion of Participants with Combined Response | Up to 96 Weeks
  Combined Response is defined as undetectable hepatitis delta virus (HDV) RNA or ≥ 2 log10 decrease in HDV RNA from baseline and normal alanine aminotransferase (ALT) normalization (ALT < upper limit of normal (ULN) at week 24).

SECONDARY OUTCOMES:
Phase 1: Proportion of Participants who Develop Antidrug Antibody (ADAs) After Administration of a Single Dose of GS-4321 and ADA Titer Characterization | First dose up to 24 Weeks
  ADA Titer characterization will include proportion of participants with ADA incidence, prevalence, persistence, and transience .
Phase 2: Serum PK Parameters AUCtau of GS-4321 | Up to 96 weeks
Phase 2: Serum PK Parameters Cmax of GS-4321 | Up to 96 Weeks
Phase 2: Serum PK Parameters Tmax of GS-4321 | Up to 96 Weeks
Phase 2: Serum PK Parameters Ctrough of GS-4321 | Up to 96 Weeks
Phase 2: Proportion of Participants With Undetectable HDV RNA or ≥ 2 log10 Decrease in HDV RNA From Baseline and normal ALT (ALT < ULN). | Weeks 4, 8, 12, 16, 20, 36, 48, 60, 72, 84, and 96
Phase 2: Change From Baseline in HDV RNA at Weeks 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, and 96 | Baseline, Weeks 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, and 96
Phase 2: Proportion of Participants With Undetectable HDV RNA | Weeks 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, and 96
Proportion of Participants With undetectable HDV RNA or ≥ 2 log10 Decrease in HDV From Baseline | Weeks 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84 and 96
Phase 2: Change From Baseline in Liver Stiffness by Elastography at Weeks 24, 48, and 96 | Weeks 24, 48, and 96
Phase 2: Proportion of Participants with normal ALT | Weeks 4, 8, 12, 16, 20, 24, 36, 48, 60, 72, 84, and 96
Phase 2: Proportion of Participants who Develop ADAs After Administration of Multiple Doses of GS-4321 and ADA Titer Characterization | First dose up to 96 Weeks plus 48 weeks of posttreatment follow-up
  ADA Titer characterization will include proportion of participants with ADA incidence, prevalence, persistence, and transience .
Phase 2: Characterize if Emergent Variants are Associated With Reduced Susceptibility to GS-4321 in Vitro and Virologic Failure in Participants With CHD | First dose up to 96 Weeks plus 48 weeks of posttreatment follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (2):
- Investigative Site, Anaheim, California, United States
- PMSI Clinical Republican Hospital "Timofei Mosneaga", Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT07096193